CLINICAL TRIAL: NCT01384747
Title: A Randomized, Double-blind Study of Effect of Fimasartan for Modification of Atheroma Vulnerability in DEFERred Coronary Disease
Brief Title: Effect of Fimasartan for Modification of Atheroma Vulnerability in DEFERred Coronary Disease (FIMA-DEFER)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVRF2011-03
Record Dates: First submitted 2011-06-24; First posted 2011-06-29 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fimasartan (Experimental): Initial dose will be started with 60mg per day. At 4 week follow-up after the procedure, dose titration upto 120 mg per day will be made if the patient is not hypotensive.
  Interventions: Drug: Fimasartan
- Placebo (Placebo Comparator): Initial dose will be started with 60mg per day. At 4 week follow-up after the procedure, dose titration upto 120 mg per day will be made if the patient is not hypotensive.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fimasartan — 60-120mg/day (target dose) of Fimasartan will be administered for the study period (till the follow-up angiography)
  Other Names: Kanarb Tab.
  Arms: Fimasartan
Drug: Placebo — 60-120mg/day (target dose) of Placebo will be administered for the study period (till the follow-up angiography)
  Arms: Placebo

SUMMARY:
* Fimasartan will be more beneficial in stabilizing the plaque vulnerability compared to control group in deferred coronary lesions.
* Fimasartan will be more beneficial in reducing total plaque volume compared to control group in deferred coronary lesions.
* Fimasartan will be more beneficial in reducing functional impairment of stenotic lesions (assessed by FFR:Fractional Flow Reserve) in deferred coronary lesions.

DETAILED DESCRIPTION:
Prospective, double-blind, randomized clinical study with enrollment of patients over at least 18 years of age who require coronary angiography for a clinical indication with hypertension defined as systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg. Inclusion requires at least one deferred coronary lesion with 1) visually-estimated angiographic %diameter stenosis 20-50% or 2) %diameter stenosis >50% without any evidence of inducible ischemia. The target vessel for IVUS interrogation must not have undergone angioplasty (deferred lesion) nor have more than 50% luminal narrowing throughout a target segment. Patients meeting inclusion criteria without any exclusion criteria will be randomized 1:1 (Fimasartan 60-120 mg vs placebo). All subjects will be followed up at 1 year for serial VH-IVUS and conventional IVUS evaluation. Also, OCT sub-study will be performed in selected patients with lesions at least 20 mm distally located from coronary ostium. All patients will be blindly assigned to control and Fimasartan once daily as 1:1 ratio and are prescribed for 1year.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertensive patients (systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg) or medically treated hypertension with normal blood pressure who undergo coronary angiography with clinical indications
2. 18 < Age < 85
3. Patient who has received informed consent
4. at least one deferred coronary lesion with 1) visually-estimated angiographic %diameter stenosis 20-50% or 2) %diameter stenosis >50% without any evidence of inducible ischemia (FFR ≥ 0.8 or negative perfusion defect on thallium scan or negative treadmill test)

Exclusion Criteria:

1. Planned cardiac surgery (e.g., CABG, valve repair or replacement, or aneurysmectomy) or planned major non-cardiac surgery within the study period
2. Planned performance of PCI or CABG in the target vessel or its branches containing the index
3. Evidence of congestive heart failure, or left ventricular ejection fraction < 40%
4. Stroke or resuscitated sudden death in the past 6 months
5. Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible)
6. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer
7. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study
8. Significant renal disease manifested by serum creatinine > 1.5 mg/dL
9. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal)
10. Active hepatitis B or C or carrier
11. Hypotension (systolic blood pressure <90 mmHg)
12. Patients already taking ACE inhibitors or ARBs
13. Patients with STEMI requiring primary PCI
14. Patients pregnant or breast-feeding or child-bearing potential
15. Patients who are lack of intention for effective contraception
16. Patients with history of previous enrollment into a clinical trials within 3 months
17. Allergic or contraindicated to Angiotensin II antagonists
18. History of any arterial bypass or angioplastic intervention involving the target vessel
19. Luminal narrowing in the left main > 50% by visual inspection of angiogram
20. Visually-estimated angiographic reference segment diameter of <2.75mm or >4.0 mm
21. Presence of thrombus or complex plaque morphology in the target vessel that suggests a high likelihood of distal embolism
22. Severe tortuosity of the target vessel or any other anatomical reasons that the investigator deems
23. Inappropriate for IVUS procedures. Vessel with thrombus (on GS-IVUS), moderate or severe calcification, angulation
24. Culprit vessel in AMI
25. RWMA (Regional Wall Motion Abnormality) or scar tissue in the territory subtended by the studied lesion

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in percent necrotic core (NC) volume of plaque by VH (Virtual Histology) in the "target segment" (within deferred vessel) | baseline and 1 year

SECONDARY OUTCOMES:
Change of total atheroma volume (TAV) and percent atheroma volume (PAV) of the target segment and the most diseased 10-mm segment (normalized to different segment length) with the largest plaque volume | baseline and 1 year
Percent change in minimal lumen area (MLA) in target segment | baseline and 1 year
Change of absolute area or percentages (%) of each plaque VH composition (fibrotic, fibrofatty, dense calcium, necrotic core) at minimal lumen area (MLA) and largest necrotic core area within the target segment | baseline and 1 year
Change of VH-IVUS (Intra Vascular UltraSound) detected plaque type from baseline | at 1 year
Change of percentage (%) of OCT (Optical Coherence Tomography)-defined TCFA (Thin Cap Fibrotic Atheroma) within the target segment from baseline | at 1 year
Change of composition of OCT-defined fibrous, fibro-calcific, and lipid-rich plaque within the target segment | baseline and 1 year
Change of OCT-defined fibrous cap thickness, the presence of plaque disruption, calcification or intraluminal thrombus within the target segment | baseline and 1 year
Change of FFR in target segment from baseline | at 1 year
systolic and diastolic blood pressure | at 1 year follow-up
Change in high sensitive CRP (C-Reactive Protein)from baseline | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Chonnam National University Hospital, Gwangju
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.